CLINICAL TRIAL: NCT01543906
Title: An Open-Label, Phase 1b, Safety/Proof-of-Concept Study to Evaluate the Effects of Oral QLT091001 in Retinitis Pigmentosa (RP) Subjects With an Autosomal Dominant Mutation in Retinal Pigment Epithelial 65 Protein (RPE65)
Brief Title: Oral QLT091001 in Retinitis Pigmentosa (RP) Subjects With an Autosomal Dominant Mutation in Retinal Pigment Epithelial 65 Protein (RPE65)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RET RP 01
Record Dates: First submitted 2012-02-17; First posted 2012-03-05 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Retinitis Pigmentosa (RP)
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — retinol acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QLT091001 (Experimental): oral QLT091001 administered once daily for 7 days
  Interventions: Drug: QLT091001

INTERVENTIONS:
Drug: QLT091001 — oral QLT091001 administered once daily for 7 days

SUMMARY:
The purpose of this study is:

* To evaluate whether 7-day treatment with oral QLT091001 can improve visual function in RP subjects with an autosomal dominant mutation in RPE65.
* To evaluate duration of visual function improvement (if observed) in RP subjects with an autosomal dominant mutation in RPE65 after 7-day treatment with oral QLT091001.
* To evaluate the safety of oral QLT091001 administered once daily for 7 days in RP subjects with an autosomal dominant mutation in RPE65.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have RP caused by an autosomal dominant mutation in RPE65, as diagnosed by an ocular geneticist or ophthalmologist.
* Subjects who have a best-corrected standard ETDRS visual acuity of 3 letters or better (20/800 Snellen equivalent) or visible photoreceptor outer segments on OCT/FAF.

Exclusion Criteria:

* Subjects with any clinically important abnormal physical finding at Screening.
* Subjects who have taken any prescription or investigational oral retinoid medication (e.g., Accutane/Roaccutane® or Soriatane/Neotigason®) within 6 months of Day 0 and subjects who did not tolerate their previous oral retinoid medication will be excluded regardless of the time of last exposure.
* Subjects with a history of diabetes or chronic hyperlipidemia, hepatitis, pancreatitis, or cirrhosis.
* Subjects who have taken any supplements containing ≥10,000 IU vitamin A within 60 days of Screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Visual field | 12 months

SECONDARY OUTCOMES:
Safety will be assessed by evaluating the following: adverse events, clinical laboratory results, ECG's and vital signs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sushanta Mallick, Study Director — QLT Inc.
Locations (2):
- Montreal Children's Hospital, McGill University Health Centre, Montreal, Quebec, Canada
- Royal Victoria Eye and Ear Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Schwartz SG, Wang X, Chavis P, Kuriyan AE, Abariga SA. Vitamin A and fish oils for preventing the progression of retinitis pigmentosa. Cochrane Database Syst Rev. 2020 Jun 18;6(6):CD008428. doi: 10.1002/14651858.CD008428.pub3. PMID 32573764